CLINICAL TRIAL: NCT04324489
Title: DAS181 for Severe COVID-19: Compassionate Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Ansun Biopharma, Inc. (Industry)
Responsible Party: Principal Investigator, Gong Zuojiong, Director, Department of Infectious Disease, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAS181-SARS-CoV-2
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; DAS181; Hypoxemia
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — oplunofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DAS181 Treatment (Experimental): Nebulized DAS181 9mg/day (4.5 mg bid/day) for 10 days
  Interventions: Drug: DAS181

INTERVENTIONS:
Drug: DAS181 — Patient receives nebulized DAS181 (4.5 mg BID/day, a total 9 mg/day) for 10 days.

SUMMARY:
The objective of the study is to investigate the safety and potential efficacy of DAS181 for the treatment of severe COVID-19.

DETAILED DESCRIPTION:
Each eligible subject is treated with DAS181 for 10 days and observed for 28 days from the first day of administration.

From day 1 to 10, once or twice a day, for 10 consecutive days, a total of 9 mg (7 ml) nebulized DAS181 is given. If DAS181 is given by twice a day, one vial containing 4.5 mg (3.5m1) DAS181 should be delivered with about 12-hour interval.

ELIGIBILITY:
Key Inclusion Criteria:

1. Positive for RNA of SARS-CoV-2 from respiratory specimens or blood specimens
2. Hypoxemic
3. Severe COVID-19
4. If female, subject must not be pregnant or nursing.
5. Non-vasectomized males are required to practice effective birth control methods
6. Capable of understanding and complying with procedures as outlined in the protocol as judged by the Investigator and able to sign informed consent form prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. ALT or AST> 8 x ULN
2. (ALT or AST> 3 x ULN) and (Total bilirubin> 2.5 x ULN or INR> 2.0 x ULN)
3. Female subjects who have a positive pregnancy test and are breastfeeding
4. Subjects using any other investigational antiviral drugs during the hospitalization before enrollment.
5. Subjects participating in other clinical trials
6. Subjects may be transferred to a non-participating hospital within 72 hours
7. People who cannot cooperate well due to mental illness, have no self-control, and cannot express clearly
8. Severe underlying diseases affecting survival
9. Critical COVID-19 requiring mechanical ventilator at the time enrolled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Improved clinical status | Day 14
  Percent of subjects with improved clinical status
Return to room air | Day 14
  Percent of subjects return to room air

SECONDARY OUTCOMES:
SARS-CoV-2 RNA | 28 days
  time to SARS-CoV-2 RNA in the respiratory specimens being undetectable
Discharge | Days 14, 21, 28
  Percent of patients discharge from hospital
Death | Day 14, 21, 28
  All-cause mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Zuojiong Gong, MD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No